CLINICAL TRIAL: NCT02271386
Title: Educating and Supporting Primary Care Providers in the Implementation of Evidence-based Practices for ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-011189
Record Dates: First submitted 2014-10-13; First posted 2014-10-22 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Evidence-Based Practice; Provider Education
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Clinicians in the intervention arm will receive the three-part intervention (Supporting Practice for ADHD, or SPA) which includes: education about ADHD management and communication training, collaborative consultation, and performance feedback, for the first 8 months of the study.
  Interventions: Behavioral: Supporting Practice for ADHD (SPA)
- Control (Other): Clinicians in the control arm will receive no intervention for the first 8 months of the study, then will receive the full SPA intervention for the last 8 months of the study.
  Interventions: Behavioral: Supporting Practice for ADHD (SPA)

INTERVENTIONS:
Behavioral: Supporting Practice for ADHD (SPA) — The SPA intervention will last for 8 months for each study arm (first 8 months of the study for the intervention group, last 8 months for the control group). The intervention includes 3 components: 1) a series of web-based educational presentations to provide education to providers about evidence-based practice for managing ADHD and strategies for promoting effective communication with families 2) Collaborative consultation designed to address clinical issues arising in practice will be provided by members of the study team.
  3) Providers will be given systematic performance feedback with regard to their use of evidence-based practices for ADHD every 2 months during the 8-month intervention period.

SUMMARY:
Although numerous studies have demonstrated that a high percentage of primary care providers (PCPs) are knowledgeable about the American Academy of Pediatrics' guidelines for managing ADHD, many fail to implement these guidelines correctly. The goal of this project is to increase the use of evidence-based practices (EBP) for assessing and treating children with ADHD between 5 and 12 years in the context of primary care practice. This randomized controlled trial will evaluate the whether a 3-part intervention (education about ADHD management and communication training, collaborative consultation, and performance feedback regarding use of EBPs) is effective in improving EBP use among primary care providers.

ELIGIBILITY:
Primary Subjects: Clinicians

Inclusion Criteria:

* Non-resident clinician (physician or nurse practitioner) at participating site

Exclusion Criteria:

* Residents

Secondary Subjects: Families

Inclusion Criteria:

* Children aged 5-12 years receiving care from a clinician enrolled in the study for ADHD and their parents

Exclusion Criteria:

* Autism spectrum disorder

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 895 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Thomas Power, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: The same group of 105 clinicians participated during both periods. Charts were reviewed for a different random sample of patients in each period (790 patients in total: 391 in the baseline and 399 in the intervention period)
Groups:
- Intervention Clinicians: Clinicians in the intervention arm received the three-part intervention (Supporting Practice for ADHD, or SPA) which includes: education about ADHD management and communication training, collaborative consultation, and performance feedback, for the first 8 months of the study.
- Control Clinicians: Clinicians in the control arm received no intervention for the first 8 months of the study, then received the full SPA intervention for the last 8 months of the study.
- Patients of Intervention Clinicians: Children aged 5-12 with ADHD seen by a clinician in the intervention group during the study period.
- Patients of Control Clinicians: Children aged 5-12 with an ADHD diagnosis seen by clinicians in the control group during the study period.
Period: Baseline Period- 8 Months
Arm/Group | Intervention Clinicians | Control Clinicians | Patients of Intervention Clinicians | Patients of Control Clinicians
Started | 53 | 52 | 200 | 191
Completed | 53 | 52 | 200 | 191
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period- 8 Months
Arm/Group | Intervention Clinicians | Control Clinicians | Patients of Intervention Clinicians | Patients of Control Clinicians
Started | 53 | 52 | 202 | 197
Completed | 53 | 52 | 202 | 197
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Clinicians | Control Clinicians | Patients of Intervention Clinicians | Patients of Control Clinicians | Total
Number analyzed (Participants) | 53 | 52 | 402 | 388 | 895
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was only measured for patients.
  years
    number analyzed (Participants) | 0 | 0 | 402 | 388 | 790
    (all) |  |  | 9.3 (1.9) | 9.2 (2.0) | 9.3 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 107 | 129 | 324
  Male | 10 | 7 | 295 | 259 | 571
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was only recorded for patients.
  Participants
    number analyzed (Participants) | 0 | 0 | 402 | 388 | 790
    Hispanic or Latino |  |  | 16 | 18 | 34
    Not Hispanic or Latino |  |  | 386 | 370 | 756
    Unknown or Not Reported |  |  | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race was only recorded for patients.
  Participants
    White: number analyzed (Participants) | 0 | 0 | 402 | 388 | 790
    White |  |  | 248 | 143 | 391
    Black: number analyzed (Participants) | 0 | 0 | 402 | 388 | 790
    Black |  |  | 104 | 221 | 325
    Other: number analyzed (Participants) | 0 | 0 | 402 | 388 | 790
    Other |  |  | 50 | 24 | 74
Insurance payer [Count of Participants; unit: Participants] — Population: Insurance payer was only recorded for patients.
  Participants
    number analyzed (Participants) | 0 | 0 | 402 | 388 | 790
    Medicaid |  |  | 169 | 224 | 393
    Private |  |  | 230 | 163 | 393
    Missing |  |  | 3 | 1 | 4
Provider Type [Count of Participants; unit: Participants] — Population: Provider type is only applicable to clinician participants.
  Participants
    number analyzed (Participants) | 53 | 52 | 0 | 0 | 105
    Pediatrician | 45 | 48 |  |  | 93
    Nurse Practitioner | 8 | 4 |  |  | 12
Baseline Perception of Acceptability of Managing ADHD in Primary Care- Assessing ADHD [Mean (Standard Deviation); unit: units on a scale] — These items are from the previously validated ADHD Questionnaire for Primary Care Providers. Scores ranged from 1 to 4, with 4 indicating the highest level of acceptability for each practice activity. Population: This measure only applies to clinicians.
  units on a scale
    number analyzed (Participants) | 53 | 52 | 0 | 0 | 105
    (all) | 3.2 (0.6) | 3.3 (0.4) |  |  | 3.3 (0.5)
Baseline Perception of Acceptability of Managing ADHD in Primary Care- Providing Mental Health Care [Mean (Standard Deviation); unit: units on a scale] — These items are from the previously validated ADHD Questionnaire for Primary Care Providers. Scores ranged from 1 to 4, with 4 indicating the highest level of acceptability for each practice activity. Population: This measure only applies to clinicians.
  units on a scale
    number analyzed (Participants) | 53 | 52 | 0 | 0 | 105
    (all) | 3.4 (0.5) | 3.4 (0.5) |  |  | 3.4 (0.5)
Baseline Perception of Acceptability of Managing ADHD in Primary Care- Recommending Medications [Mean (Standard Deviation); unit: units on a scale] — These items are from the previously validated ADHD Questionnaire for Primary Care Providers. Scores ranged from 1 to 4, with 4 indicating the highest level of acceptability for each practice activity. Population: This measure only applied to clinicians.
  units on a scale
    number analyzed (Participants) | 53 | 52 | 0 | 0 | 105
    (all) | 3.5 (0.6) | 3.6 (0.4) |  |  | 3.6 (0.5)
Perceived effectiveness at managing ADHD in primary care [Mean (Standard Deviation); unit: units on a scale] — These items are from the previously validated ADHD Questionnaire for Primary Care Providers. Scores ranged from 1 to 4, with 4 indicating the highest level of acceptability for each practice activity. Population: This measure only applies to clinicians.
  units on a scale
    number analyzed (Participants) | 53 | 52 | 0 | 0 | 105
    (all) | 2.9 (0.8) | 3.1 (0.6) |  |  | 3.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Were Sent the Parents Rating Scale
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a parent rating scale was sent out during the baseline interval
Time Frame: Baseline Period (8 months)
Population: We reviewed charts for a total of 402 patients of intervention clinicians (200 who had an office visit in the 8-month baseline period and 202 who had an office visit in the 8-month intervention period). We reviewed charts for a total of 388 patients of control clinicians (191 in the baseline period and 197 in the control period).
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 200 | 191
Participants | 33 | 37

2. Primary Outcome: Number of Patients Whose Parent Rating Scale Was Returned
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a parent rating scale was received by the clinician during the baseline interval
Time Frame: Baseline Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 200 | 191
Participants | 29 | 28

3. Primary Outcome: Number of Patients Who Were Sent the Teacher Rating Scale
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a teacher rating scale was sent out during the baseline interval
Time Frame: Baseline Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 200 | 191
Participants | 33 | 34

4. Primary Outcome: Number of Patients Whose Teacher Rating Scale Was Returned
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a teacher rating scale was received by the clinician during the baseline interval
Time Frame: Baseline Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 200 | 191
Participants | 28 | 31

5. Primary Outcome: Number of Patients Who Were Sent the Parents Rating Scale
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a parent rating scale was sent out during the intervention interval
Time Frame: Intervention Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 202 | 197
Participants | 85 | 65

6. Primary Outcome: Number of Patients Whose Parent Rating Scale Was Returned
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a parent rating scale was received by the clinician during the intervention interval
Time Frame: Intervention Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 202 | 197
Participants | 59 | 47

7. Primary Outcome: Number of Patients Who Were Sent the Teacher Rating Scale
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a teacher rating scale was sent out during the intervention interval
Time Frame: Intervention Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 202 | 197
Participants | 67 | 60

8. Primary Outcome: Number of Patients Whose Teacher Rating Scale Was Returned
Description: This measure is based on chart review of patients of clinicians in each study arm (up to 4 patients per clinician) and reflects whether there is evidence that a teacher rating scale was received by the clinician during the intervention interval
Time Frame: Intervention Period (8 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians | Patients of Control Clinicians
Number analyzed (Participants) | 202 | 197
Participants | 52 | 47

9. Secondary Outcome: Number of Patients Who Were Sent the Parent Rating Scale - by MOC Status
Description: We calculated the percent of patient charts with evidence that a parent rating scale was sent out during the baseline period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Baseline Period (8 months)
Population: This outcome was only assessed for patients of clinicians in the intervention group, and compared patients of clinicians who did and did not fulfill all requirements to receive Maintenance of Certification (MOC) credit. The MOC group included 76 patients in the baseline and 73 in the intervention period. The non-MOC group included 124 and 129.
Measure: Count of Participants; unit: Participants
Groups:
- Patients of Intervention Clinicians Completing MOC Attestation: Children aged 5-12 with ADHD seen by a clinician in the intervention group who fulfilled all requirements to receive Maintenance of Certification (MOC) credit.
- Patients of Intervention Clinicians Not Completing MOC Attesta: Children aged 5-12 with ADHD seen by a clinician in the intervention group who did not fulfill all requirements to receive Maintenance of Certification (MOC) credit.
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 76 | 124
Participants | 12 | 21

10. Secondary Outcome: Number of Patients Whose Parent Rating Scale Was Returned- by MOC Status
Description: We calculated the percent of patient charts with evidence that a parent rating scale was received by the clinician/practice during the baseline period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Baseline Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 76 | 124
Participants | 12 | 17

11. Secondary Outcome: Number of Patients Who Were Sent the Teacher Rating Scale- by MOC Status
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was sent out during the baseline period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Baseline Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 76 | 124
Participants | 12 | 21

12. Secondary Outcome: Number of Patients Whose Teacher Rating Scale Was Returned- by MOC Status
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was received by the clinician/practice during the baseline period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Baseline Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 76 | 124
Participants | 12 | 16

13. Secondary Outcome: Number of Patients Who Were Sent the Parent Rating Scale- by MOC Status
Description: We calculated the percent of patient charts with evidence that a parent rating scale was sent out during the intervention period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Intervention Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 73 | 129
Participants | 40 | 45

14. Secondary Outcome: Number of Patients Whose Parent Rating Scale Was Returned- by MOC Status
Description: We calculated the percent of patient charts with evidence that a parent rating scale was received by the clinician/practice during the intervention period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Intervention Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 73 | 129
Participants | 26 | 33

15. Secondary Outcome: Number of Patients Who Were Sent the Teacher Rating Scale- by MOC Status
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was sent out during the intervention period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Intervention Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 73 | 129
Participants | 28 | 39

16. Secondary Outcome: Number of Patients Whose Teacher Rating Scale Was Returned- by MOC Status
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was received by the clinician/practice during the intervention period, separately for intervention clinicians who did and did not complete Maintenance of Certification (MOC) attestation.
Time Frame: Intervention Period (8 months)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Completing MOC Attestation | Patients of Intervention Clinicians Not Completing MOC Attesta
Number analyzed (Participants) | 73 | 129
Participants | 21 | 31

17. Secondary Outcome: Number of Patients Who Were Sent the Parent Rating Scale- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a parent rating scale was sent out during the baseline period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Baseline Period (8 months)
Population: This outcome was only assessed for patients of clinicians in the intervention group, and compared patients of clinicians who did and did not participate in at least one performance feedback call. The feedback call group included 115 patients in the baseline and 112 in the intervention period. The non-feedback call group included 85 and 90.
Measure: Count of Participants; unit: Participants
Groups:
- Patients of Intervention Clinicians Participating in >=1 Call: Children aged 5-12 with ADHD seen by a clinician in the intervention group who participated in at least one performance feedback call.
- Patients of Intervention Clinicians Participating in 0 Calls: Children aged 5-12 with ADHD seen by a clinician in the intervention group who did not participate in at least one performance feedback call.
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 115 | 85
Participants | 21 | 12

18. Secondary Outcome: Number of Patients Whose Parent Rating Scale Was Returned- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a parent rating scale was received by the clinician/practice during the baseline period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Baseline Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 115 | 85
Participants | 19 | 10

19. Secondary Outcome: Number of Patients Who Were Sent the Teacher Rating Scale- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was sent out during the baseline period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Baseline Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 115 | 85
Participants | 24 | 9

20. Secondary Outcome: Number of Patients Whose Teacher Rating Scale Was Returned- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was received by the clinician/practice during the baseline period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Baseline Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 115 | 85
Participants | 21 | 7

21. Secondary Outcome: Number of Patients Who Were Sent the Parent Rating Scale- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a parent rating scale was sent out during the intervention period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Intervention Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 112 | 90
Participants | 56 | 29

22. Secondary Outcome: Number of Patients Whose Parent Rating Scale Was Returned- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a parent rating scale was received by the clinician/practice during the intervention period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Intervention Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 112 | 90
Participants | 35 | 24

23. Secondary Outcome: Number of Patients Who Were Sent the Teacher Rating Scale- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was sent out during the intervention period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Intervention Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 112 | 90
Participants | 42 | 25

24. Secondary Outcome: Number of Patients Whose Teacher Rating Scale Was Returned- by Feedback Call Participation
Description: We calculated the percent of patient charts with evidence that a teacher rating scale was received by the clinician/practice during the intervention period, separately for intervention clinicians who did and did not participate in at least one performance feedback call.
Time Frame: Intervention Period (8 months)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Intervention Clinicians Participating in >=1 Call | Patients of Intervention Clinicians Participating in 0 Calls
Number analyzed (Participants) | 112 | 90
Participants | 30 | 22

25. Secondary Outcome: Implementation Outcome: Number of Clinicians Who Completed All 3 Educational Presentations
Description: We assessed the proportion of clinicians randomized to the intervention group that completed all 3 educational presentations.
Time Frame: Intervention Period (8 months)
Population: This outcome was only assessed for intervention clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Clinicians | Control Clinicians
Number analyzed (Participants) | 53 | 0
Participants | 42 |

26. Secondary Outcome: Implementation Outcome: Number of Clinicians Who Used the Collaborative Consultation Component
Description: We calculated the proportion of clinicians in the intervention group that posted in the online networking site which was used to facilitate collaborative consultation.
Time Frame: Intervention Period (8 months)
Population: This outcome was only assessed for intervention clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Clinicians | Control Clinicians
Number analyzed (Participants) | 53 | 0
Participants | 5 |

27. Secondary Outcome: Implementation Outcome: Number of Clinicians Who Participated in at Least One Performance Feedback Call
Description: We calculated the proportion of clinicians in the intervention group who participated in at least one of the four performance feedback calls that were held during the study period.
Time Frame: Intervention Period (8 months)
Population: This outcome was only assessed for intervention clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Clinicians | Control Clinicians
Number analyzed (Participants) | 53 | 0
Participants | 30 |

28. Secondary Outcome: Implementation Outcome: Number of Clinicians Who Participated in All Intervention Components and Attested to Fulfilling MOC Requirements
Description: We calculated the proportion of clinicians in the intervention group who completed all components of the intervention and attested to fulfilling MOC requirements.
Time Frame: Intervention Period (8 months)
Population: This outcome was only assessed for intervention clinicians.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Clinicians | Control Clinicians
Number analyzed (Participants) | 53 | 0
Participants | 19 |

ADVERSE EVENTS:
Time Frame: 16 months (8 month baseline period and 8 month intervention period)
Arm/Group | Intervention Clinicians | Control Clinicians | Patients of Intervention Clinicians | Patients of Control Clinicians
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52 | 0/402 | 0/388
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/402 | 0/388
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/402 | 0/388

LIMITATIONS AND CAVEATS:
Enrollment occurred within 1 health system among clinicians who were interested in participating in the project and worked in practices that agreed to participate, which may limit generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No